CLINICAL TRIAL: NCT02768129
Title: tDCS for Chronic Low Back Pain: A Study Examining the Effect of Transcranial Direct Current Stimulation on the Emotional Response to Chronic Low Back Pain
Brief Title: Transcranial Direct Current Stimulation for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1411-003
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- sham tDCS (Sham Comparator): 10 sessions sham transcranial direct current stimulation (tDCS)
  Interventions: Device: sham transcranial direct current stimulation
- active tDCS (Experimental): 10 sessions active transcranial direct current stimulation (tDCS)
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — active stimulation: 2 milliamp (mA), 20 mins
  Arms: active tDCS
Device: sham transcranial direct current stimulation — sham stimulation
  Arms: sham tDCS

SUMMARY:
The goal of this study is to investigate the role of central neural pathways in mediating chronic pain. The aim of the study is to test the effect of stimulating brain regions that are part of a network underlying central pain processing using a non-invasive brain stimulation technique, transcranial Direct Current Stimulation (tDCS). Prior studies have used tDCS to target both sensory related cortical areas and those important for higher-order representations of pain. This study will target brain regions important for the behavioral response to the chronic sensation of pain. The hypothesis is that stimulation of these brain regions can modulate not only the affective component of pain, but ultimately also improve functioning and quality of life. This hypothesis will be tested by treating study participants eighteen and older with chronic low back pain (CLBP) of greater than six months using tDCS. To be part of this study, participants must meet all the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low Back Pain ≥ 6 months duration in the lumbar region, present more than half the days of the month, and on average be at a moderate level of severity in the last month
* At least one trial of physician recommended medication (e.g. acetaminophen, NSAIDS, skeletal muscle relaxants)
* Pre-existing opioid and non-opioid pain medication must be non-existent or stable (medications have not changed for one month)
* Be able to understand, read and write English
* If female and of childbearing age, agree to use acceptable birth control during the study treatment period (oral contraceptives, history of tubal ligation, history of a hysterectomy, or a reliable barrier method)

Exclusion Criteria:

* Lifetime Diagnostic and Statistical Manual (DSM) IV diagnosis of bipolar disorder, schizophrenia, or other chronic psychotic condition
* Current DSM-IV diagnosis of substance dependence for alcohol, sedative/hypnotic drugs, stimulants, cocaine
* Current cancer, infection, or inflammatory arthritis
* Broken skin or other lesions in the area of the electrodes
* Uncontrolled medical problems, such as diabetes mellitus, hypertension, pulmonary or airway disease, heart failure, coronary artery disease, or any other condition that poses a risk for the subject during participation
* Presence of metal in the cranial cavity
* Holes in the skull made by trauma or surgery
* Pacemakers, medication pumps, and other implanted electronic hardware
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 30 participants that were consented, 9 participants were ineligible, withdrew, or were lost to contact before commencing tDCS.
Groups:
- Sham tDCS: 10 sessions sham transcranial direct current stimulation (tDCS)
  sham transcranial direct current stimulation: sham
Period: Overall Study
Arm/Group | Sham tDCS | Active tDCS
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The data collected from the 21 participants who completed tDCS treatment (either active or sham) is included in the analysis.
Groups:
- Active tDCS: 10 sessions sham transcranial direct current stimulation (tDCS)
  sham transcranial direct current stimulation: active : 2 mA, 20 mins
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.8) | 60.7 (11.8) | 63.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 7 | 14
  Black or African American | 0 | 1 | 1
  Hispanic or Latino | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 2 | 3 | 5
Years of Education [Mean (Standard Deviation); unit: years] | 14.0 (2.6) | 14.7 (2.6) | 14.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: West Haven-Yale Multidimensional Pain Inventory (General Activity Subscale) Rating
Description: Subscale C of the West Haven-Yale Multidimensional Pain Inventory (WHY-MPI) is a validated measure of chronic pain's effects on functioning. Ranging from 0-108, higher scores indicate more activity (better outcome).
Time Frame: 8 weeks total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 11 | 10
score on a scale | 35.3 (17.7) | 48.4 (21.2)

2. Primary Outcome: Pain Anxiety Symptom Scale Rating
Description: The Pain Anxiety Symptom Scale (PASS-20) is a validated measure of pain-related avoidance and fear. Total score ranges 0-100. Higher scores indicate greater pain anxiety.
Time Frame: 8 weeks total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 11 | 10
score on a scale | 26.4 (22.0) | 26.3 (23.6)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Sham tDCS | Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
small sample (N=21), participants not stratified by premorbid anxiety levels, inability to guarantee optimal targeting of left dorsal anterior cingulate cortex (dACC) in all participants, inability to address laterality effects of pain perception

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT02768129/Prot_SAP_000.pdf